CLINICAL TRIAL: NCT00156715
Title: Efficacy of Quetiapine in Treating Patients With Active Substance Use Disorder and Schizophrenia
Brief Title: Efficacy of Quetiapine in the Treatment of Patients With Schizophrenia and a Comorbid Substance Use Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Augusta University (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Alan Green, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16563; IRUSQUET0063 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2005-09-06; First posted 2005-09-12 (Estimated); Results first posted 2010-12-21 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychotic Disorder; Substance Abuse; Alcohol Abuse
Keywords: Quetiapine; Seroquel; Schizophrenia; Dual Diagnosis; Substance Abuse; Alcohol Abuse
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Substance-Related Disorders; Alcoholism | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quetiapine (Experimental): After patients provided informed consent and completed baseline measures, quetiapine was initiated in all participants and titrated up to a target dose of 600 mg (in divided daily doses) over two weeks as the previous antipsychotic medication was slowly tapered and discontinued. Participants met with study physicians weekly to assess tolerability and response to the medication. Concomitant medications were held constant. After the initial titration period, quetiapine was dosed in a flexible manner up to 800 mg /day, with dose adjustments based on symptomatic response and side effects.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — After patients provided informed consent and completed baseline measures, quetiapine was initiated in all participants and titrated up to a target dose of 600 mg (in divided daily doses) over two weeks as the previous antipsychotic medication was slowly tapered and discontinued. Participants met with study physicians weekly to assess tolerability and response to the medication. Concomitant medications were held constant. After the initial titration period, quetiapine was dosed in a flexible manner up to 800 mg /day, with dose adjustments based on symptomatic response and side effects.
  Other Names: Seroquel

SUMMARY:
The purpose of this study is to examine the efficacy of quetiapine (Seroquel) in reducing substance use in persons diagnosed with schizophrenia. The primary hypothesis is that quetiapine treatment will be associated with a decrease in substance use.

DETAILED DESCRIPTION:
Comorbid alcohol/substance use disorder (SUD) in schizophrenia is a major concern, both in view of the high frequency of SUD among patients with schizophrenia and the difficulty in managing such patients. Though antipsychotic medications are effective in reducing symptoms and impairment in persons with schizophrenia, the typical antipsychotic agents are of limited value in controlling alcohol/substance use in these patients. Extrapyramidal, dysphoric side effects of conventional neuroleptics may actually promote the use of substances in an attempt to counteract these effects.

Novel antipsychotics have radically altered treatment expectations and outcomes for patients with severe forms of schizophrenia. With the greater availability of novel agents in clinical practice, it has been noted that these benefits have also extended to specific subgroups of patients including patients with comorbid SUD. Several retrospective studies have demonstrated a decrease in comorbid substance use in patients with schizophrenia treated with clozapine. There is little data available, however, on the efficacy of quetiapine in patients with schizophrenia and comorbid SUD. Its receptor profile, including a weak Dopamine2 (D2) receptor blocking ability and substantial effects at noradrenergic receptors, makes it a logical antipsychotic to use in the comorbid population.

The study is an open-label investigation of the efficacy of quetiapine in a group of 30 patients with schizophrenia and comorbid substance use disorder. Patients diagnosed with schizophrenia or schizoaffective disorder and a comorbid substance use disorder are switched to quetiapine for 12 weeks. We hypothesize that quetiapine treatment will be associated with a decrease in substance use. Moreover, we further hypothesize that measures of symptoms, cognition and quality of life will also improve over baseline assessments in patients treated with quetiapine. Data suggesting a beneficial effect of quetiapine will have to be confirmed in a prospective double-blind study. This pilot investigation will provide preliminary data and effect sizes that will be used in the design of this subsequent investigation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Schizophrenia or schizoaffective disorder
* Meets Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (SCID) criteria for a substance use disorder (alcohol use disorder [AUD]; abuse or dependence)
* Active substance use on at least 8 days during the 4 weeks prior to randomization.
* Current treatment with antipsychotic medication.
* Able to provide informed consent, or in the case of patients with legal court appointed guardians willing to give assent, with the consent of the guardian.
* Not actively suicidal.

Exclusion Criteria:

* Current treatment with, decanoate antipsychotic, clozapine, or doses of quetiapine not approved by the team of investigators. Individuals treated with depot antipsychotic must wait until the end of their injection cycle before starting on study medication.
* Currently pregnant, planning to become pregnant, or unwilling to use an acceptable form of birth control.
* Currently residing in a residential program designed to treat substance use disorders.
* Treatment at baseline with a psychotropic agent proposed to curtail substance use.
* Patients who, in the opinion of the investigator, are judged unsuitable to participate in the study.
* Unable to take part in the assessments in a meaningful way
* Hypersensitivity/intolerance to quetiapine
* Serious, unstable medical condition
* Participation in clinical trial of an investigational drug within 30 days of baseline visit, or concurrent participation in a treatment study of a psychosocial intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-03; Primary Completion 2006-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan I Green, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - Medical College of Georgia, Augusta, Georgia
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - West Central Behavioral Health, Lebanon, New Hampshire
  - Mental Health Center of Greater Manchester, Manchester, New Hampshire

REFERENCES:
- [Background] Albanese MJ, Khantzian EJ, Murphy SL, Green AI. Decreased substance use in chronically psychotic patients treated with clozapine. Am J Psychiatry. 1994 May;151(5):780-1. doi: 10.1176/ajp.151.5.780b. No abstract available. PMID 8166327
- [Background] Bartels SJ, Teague GB, Drake RE, Clark RE, Bush PW, Noordsy DL. Substance abuse in schizophrenia: service utilization and costs. J Nerv Ment Dis. 1993 Apr;181(4):227-32. doi: 10.1097/00005053-199304000-00003. PMID 8473874
- [Background] Bowers MB Jr, Mazure CM, Nelson JC, Jatlow PI. Psychotogenic drug use and neuroleptic response. Schizophr Bull. 1990;16(1):81-5. doi: 10.1093/schbul/16.1.81. PMID 1970670
- [Background] Brown ES, Nejtek VA, Perantie DC, Rajan Thomas N, Rush AJ. Cocaine and amphetamine use in patients with psychiatric illness: a randomized trial of typical antipsychotic continuation or discontinuation. J Clin Psychopharmacol. 2003 Aug;23(4):384-8. doi: 10.1097/01.jcp.0000085412.08426.08. PMID 12920415
- [Background] Buckley PF, Naber D: Quetiapine and sertindole: clinical use and experience. In: Schizophrenia and Mood Disorders: The New Drug Therapies in Clinical Practice. Edited by PF Buckley and JL Waddington. Butterworth-Heinemann, 2000.
- [Background] Buckley P, Thompson PA, Way L, Meltzer HY. Substance abuse and clozapine treatment. J Clin Psychiatry. 1994 Sep;55 Suppl B:114-6. PMID 7961553
- [Background] Buckley PF. Novel antipsychotic medications and the treatment of comorbid substance abuse in schizophrenia. J Subst Abuse Treat. 1998 Mar-Apr;15(2):113-6. doi: 10.1016/s0740-5472(97)00134-7. PMID 9561949
- [Background] Buckley PF. Substance abuse in schizophrenia: a review. J Clin Psychiatry. 1998;59 Suppl 3:26-30. PMID 9541335
- [Background] Buckley PF, Miller A, Chiles JA, Sajatovic M. Implementing effectiveness research and improving care for schizophrenia in real-world settings. Am J Manag Care. 1999 Jun 25;5 Spec No:SP47-56. PMID 10538860
- [Background] Buckley P, McCarthy M, Chapman P, Richman C, Yamamoto B. Clozapine treatment of comorbid substance abuse in patients with schizophrenia. Schizophr Res 1999; 36: 272.
- [Background] Carey KB, Cocco KM, Simons JS. Concurrent validity of clinicians' ratings of substance abuse among psychiatric outpatients. Psychiatr Serv. 1996 Aug;47(8):842-7. doi: 10.1176/ps.47.8.842. PMID 8837156
- [Background] Conley RR, Kelly DL, Gale EA. Olanzapine response in treatment-refractory schizophrenic patients with a history of substance abuse. Schizophr Res. 1998 Sep 7;33(1-2):95-101. doi: 10.1016/s0920-9964(98)00062-0. PMID 9783349
- [Background] Drake RE, Osher FC, Noordsy DL, Hurlbut SC, Teague GB, Beaudett MS. Diagnosis of alcohol use disorders in schizophrenia. Schizophr Bull. 1990;16(1):57-67. doi: 10.1093/schbul/16.1.57. PMID 2333482
- [Background] Drake RE, Xie H, McHugo GJ, Green AI. The effects of clozapine on alcohol and drug use disorders among patients with schizophrenia. Schizophr Bull. 2000;26(2):441-9. doi: 10.1093/oxfordjournals.schbul.a033464. PMID 10885642
- [Background] Green AI, Alam MY, Sobieraj JT, Pappalardo KM, Waternaux C, Salzman C, Schatzberg AF, Schildkraut JJ. Clozapine response and plasma catecholamines and their metabolites. Psychiatry Res. 1993 Feb;46(2):139-49. doi: 10.1016/0165-1781(93)90016-a. PMID 8483973
- [Background] Green AI, Alam MY, Boshes RA, Waternaux C, Pappalardo KM, Fitzgibbon ME, Tsuang MT, Schildkraut JJ. Haloperidol response and plasma catecholamines and their metabolites. Schizophr Res. 1993 Jun;10(1):33-7. doi: 10.1016/0920-9964(93)90074-s. PMID 8369230
- [Background] Green AI, Zimmet SV, Strous RD, Schildkraut JJ. Clozapine for comorbid substance use disorder and schizophrenia: do patients with schizophrenia have a reward-deficiency syndrome that can be ameliorated by clozapine? Harv Rev Psychiatry. 1999 Mar-Apr;6(6):287-96. doi: 10.3109/10673229909017206. PMID 10370435
- [Background] Heinrichs DW, Hanlon TE, Carpenter WT Jr. The Quality of Life Scale: an instrument for rating the schizophrenic deficit syndrome. Schizophr Bull. 1984;10(3):388-98. doi: 10.1093/schbul/10.3.388. PMID 6474101
- [Background] Khantzian EJ. The self-medication hypothesis of addictive disorders: focus on heroin and cocaine dependence. Am J Psychiatry. 1985 Nov;142(11):1259-64. doi: 10.1176/ajp.142.11.1259. PMID 3904487
- [Background] Khantzian EJ. The self-medication hypothesis of substance use disorders: a reconsideration and recent applications. Harv Rev Psychiatry. 1997 Jan-Feb;4(5):231-44. doi: 10.3109/10673229709030550. PMID 9385000
- [Background] Meats P. Quetiapine ('Seroquel'); an effective and well-tolerated atypical antipsychotic. Int J Psychiatry Clin Pract. 1997;1(4):231-9. doi: 10.3109/13651509709024734. PMID 24946189
- [Background] Siris SG. Pharmacological treatment of substance-abusing schizophrenic patients. Schizophr Bull. 1990;16(1):111-22. doi: 10.1093/schbul/16.1.111. PMID 1970669
- [Background] Small JG, Hirsch SR, Arvanitis LA, Miller BG, Link CG. Quetiapine in patients with schizophrenia. A high- and low-dose double-blind comparison with placebo. Seroquel Study Group. Arch Gen Psychiatry. 1997 Jun;54(6):549-57. doi: 10.1001/archpsyc.1997.01830180067009. PMID 9193196
- [Background] Zimmet SV, Strous RD, Burgess ES, Kohnstamm S, Green AI. Effects of clozapine on substance use in patients with schizophrenia and schizoaffective disorder: a retrospective survey. J Clin Psychopharmacol. 2000 Feb;20(1):94-8. doi: 10.1097/00004714-200002000-00016. PMID 10653215
- [Background] Arvanitis LA, Miller BG. Multiple fixed doses of "Seroquel" (quetiapine) in patients with acute exacerbation of schizophrenia: a comparison with haloperidol and placebo. The Seroquel Trial 13 Study Group. Biol Psychiatry. 1997 Aug 15;42(4):233-46. doi: 10.1016/s0006-3223(97)00190-x. PMID 9270900
- [Background] Weiden PJ. Quetiapine ('seroquel'): a new 'atypical' antipsychotic. J Prac Psychiatry and Behav Health 1997; 3(6): 368-374.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two urban study sites, one in New England, the other in the Southeast, primarily through clinician referral, over two years. All participants gave informed consent.
Pre-assignment Details: Prior to starting quetiapine, all participants first completed a screening assessment to establish diagnosis, amount of alcohol (and other drugs) consumed, and current medications and medical status. This data was used to characterize the group and assess whether they met eligibility criteria for the study.
Groups:
- QUET: After patients provided informed consent and completed baseline measures, quetiapine was initiated in all participants and titrated up to a target dose of 600 mg (in divided daily doses) over two weeks as the previous antipsychotic medication was slowly tapered and discontinued. Participants met with study physicians weekly to assess tolerability and response to the medication. Concomitant medications were held constant. After the initial titration period, quetiapine was dosed in a flexible manner up to 800 mg /day, with dose adjustments based on symptomatic response and side effects.
Period: Overall Study
Arm/Group | QUET
Started | 23
Completed | 16
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | QUET
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Drinking Days Per Week
Description: Timeline Follow-back (TLFB) procedure was used at screening and baseline to establish current substance use, and it was also used weekly during the course of the study to assess continued alcohol and other substance use. TLFB cosisted of using a calendar and sasking participants to report alcohol and other drug use since last visit. At the screening visit, the TLFB was done for the four weeks prior to the visit.
Time Frame: 12 Weeks
Population: Only those participants who received at least 4 weeks of treatment with quetiapine were included in this analysis. Site differences resulted in only the 11 participants from Site 1 to be included in the analysis. Participants from Site 2 were all admitted to the study directly from the hospital which could have affected their alcohol consumption.
Measure: Mean (Standard Deviation); unit: Drinking Days per Week
Arm/Group | QUET
Number analyzed (Participants) | 11
Drinking Days per Week | 2.7 (2.3)

2. Secondary Outcome: Clinical Symptoms
Description: The main outcome measure of clinical symptoms was the Positive and Negative Symptoms Scale. This is a 30 item scale for assessing patients diagnosed with schizophrenia. Each item is rated on a 1 (absent) to 7 (extreme) scale. The minimum total score is 30 and the maximum is 210.
Time Frame: 12 Weeks
Population: Only those participants who received at least 4 weeks of treatment with quetiapine were included in this analysis. Site differences resulted in only the 11 participants from Site 1 to be included in this analysis. Participants from Site 2 were all admitted to the study directly from the hospital, which could have affected their behavior.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | QUET
Number analyzed (Participants) | 11
Units on a scale | 65.5 (16.5)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | QUET
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QUET (N=16)
Increased Psychosis (Psychiatric disorders) | 2 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lump in Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Could not obtain biopsy results
Suicidal Ideation/Attempt (Psychiatric disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QUET (N=16)
Dry Mouth (General disorders) | 7 (7)
Sleeplessness (General disorders) | 4 (4)
Pain (General disorders) | 3 (3)
Increased Appetite/Weight Gain (Metabolism and nutrition disorders) | 5 (5)
Gi Distress/Poor Appetite (Gastrointestinal disorders) | 2 (2)
Cold or Flu Symptoms (General disorders) | 4 (5)
Sedation (General disorders) | 7 (9)
Unusual Dream Activity (Psychiatric disorders) | 3 (3)
Heaviness/Pressure (General disorders) | 2 (2)
Dizzy (General disorders) | 3 (3)
Hypertension (Cardiac disorders) | 2 (2)
Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Palpatations (Cardiac disorders) | 1 (1)
Other (General disorders) | 4 (7)

LIMITATIONS AND CAVEATS:
Lack of a control group; Small study group size, and the consequent lack of power to detect a significant change; Differences between the populations at the two sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No